CLINICAL TRIAL: NCT02707965
Title: Characterization of Epilepsy Patients At-risk for Adverse Outcomes Related to Switching Antiepileptic Drug Products: BEEP 2b Study
Brief Title: Characterization of Epilepsy Patients BEEP 2b
Acronym: BEEP2b
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-107D; HHSF223201400188C (Other Grant/Funding Number: USFDA)
Record Dates: First submitted 2016-02-26; First posted 2016-03-14 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Epilepsy
Keywords: Generic brittle; Anti-epileptic drug; Bioequivalence
MeSH Terms: conditions — Epilepsy | interventions — Oxcarbazepine; Valproic Acid; Carbamazepine; Lamotrigine; Levetiracetam; Topiramate; Zonisamide; Phenytoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Active Comparator): This is a crossover study with 4 treatment periods consisting of 2 Test periods(generic drug) and 2 Reference periods (brand name drug). Each treatment period lasts about 2 weeks, and patients will be randomized into one of the two sequences. All drugs are administered orally, and dosage will depend on a patient.
  Interventions: Drug: Oxcarbazepine (brand name vs generic drugs); Drug: Divalproex Sodium (brand name vs generic drugs); Drug: Carbamazepine (brand name vs generic drugs); Drug: Lamotrigine (brand name vs generic drugs); Drug: levetiracetam (brand name vs generic drugs); Drug: Topiramate (brand name vs generic drugs); Drug: Zonisamide (brand name vs generic drugs); Drug: Phenytoin sodium (brand name vs generic drugs)
- Sequence 2 (Active Comparator): This is a crossover study with 4 treatment periods consisting of 2 Test periods(generic drug) and 2 Reference periods (brand name drug). Each treatment period lasts about 2 weeks, and patients will be randomized into one of the two sequences. All drugs are administered orally, and dosage will depend on a patient.
  Interventions: Drug: Oxcarbazepine (brand name vs generic drugs); Drug: Divalproex Sodium (brand name vs generic drugs); Drug: Carbamazepine (brand name vs generic drugs); Drug: Lamotrigine (brand name vs generic drugs); Drug: levetiracetam (brand name vs generic drugs); Drug: Topiramate (brand name vs generic drugs); Drug: Zonisamide (brand name vs generic drugs); Drug: Phenytoin sodium (brand name vs generic drugs)

INTERVENTIONS:
Drug: Oxcarbazepine (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.
Drug: Divalproex Sodium (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.
Drug: Carbamazepine (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.
Drug: Lamotrigine (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.
Drug: levetiracetam (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.
Drug: Topiramate (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.
Drug: Zonisamide (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.
Drug: Phenytoin sodium (brand name vs generic drugs) — This is a cross-over replicate study with 2 sequences (arms) comparing brand name and generic anti-epileptic drugs. Subjects will take a brand name and a generic drug of the same intervention. While there are only 2 sequences, there are 8 possible drugs for this study, and a study patient will only take 1 out of 8 study drugs. Only pharmacists will know which sequence each patient is assigned to.

SUMMARY:
Some epilepsy patients are described as GB when they have worsened seizures or side effects related to switching between brand name and generic, or between generic antiepileptic drug (AED) products. In concert with Aim 1 (protocol BEEP2a), this study will uncover possible reasons for patient problems with the drug switching. Factors that will be studied in GB epilepsy patients include physiologic, psychological, and genetic factors, including in this protocol whether brand and generic AEDs are pharmacokinetically similar in GB individuals.

DETAILED DESCRIPTION:
This pilot study is exploratory research to characterize the "generic brittle" (GB) patient and to identify major causes for generic brittleness in epilepsy patients who are sensitive to antiepileptic drug (AED) formulation changes.

The primary aim of this BEEP2b study is to perform individual pharmacokinetic (PK) similarity testing of brand and generic AEDs in "probably GB" patients (N=12),who were selected on the basis of having GB-defining factors from the BEEP2a study, in order to confirm whether these factors are predictive of a generic brittle response to product switching. The study design involves a randomized, double-blind, multiple-dose, complete four-way replicate crossover design in which one brand and one generic will be compared in each patient from the patient's own AED regimen. Associated adverse events (i.e. seizures and side effects) will also be assessed. Bioequivalence (BE) will not be assessed. Rather, about nine AEDs are expected to be collectively evaluated. Generic brittleness anticipates that, for individual subjects, brand and generic may be the same or different, depending upon the underlying basis for generic brittleness. This exploratory research is focused on understanding individual patient attributes that contribute to GB, and is not focused on either product development or comparison of specific products.

ELIGIBILITY:
Inclusion Criteria:

1. Subject previously completed BEEP2a study, found to be probably GB, and able to provide informed consent or subject's legally authorized representative is able to provide informed consent.
2. Subject is male or female between 18 and 76 years of age inclusive.
3. Subject has a diagnosis of epilepsy including focal or primary generalized epilepsy.
4. Subject is taking at least one study antiepileptic drug for the treatment of epilepsy.
5. Subject is an acceptable candidate for venipuncture.
6. Subject is willing to be switched between brand and generic drug.
7. Subject is willing to stop all non-routine OTC medications for 24 hours prior to and during pharmacokinetic study visits.
8. Subject is willing to maintain stable doses of all other AEDs, including Vagus Nerve Stimulation parameters for the duration of the study.

Exclusion Criteria:

1. Subject has any medical condition, including a progressive neurological condition, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in the trial.
2. Subject has a history of alcohol or drug abuse, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in this trial.
3. Subject has a history of previous or current significant psychiatric disorder that would interfere with conduct of the study.
4. Subject is pregnant or lactating.
5. Subject has severe liver impairment as assessed by alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels ≥10 times the upper limit of normal (ULN).
6. Subject has severe renal impairment as assessed by creatinine clearance lower than 30mL/min, using the Cockcroft-Gault formula.
7. Female subjects of childbearing potential will not be eligible to participate who are unwilling or unable to use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: condom with spermicide, diaphragm with spermicide, IUD without progesterone, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence.
8. Subject is not willing or able to be adherent to study protocol (e.g. study medication dosing and any interacting comedication).

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Polli, Ph.D, Principal Investigator — University of Maryland School of Pharmacy
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- [Background] Andermann F, Duh MS, Gosselin A, Paradis PE. Compulsory generic switching of antiepileptic drugs: high switchback rates to branded compounds compared with other drug classes. Epilepsia. 2007 Mar;48(3):464-9. doi: 10.1111/j.1528-1167.2007.01007.x. PMID 17346246
- [Background] Zachry WM 3rd, Doan QD, Clewell JD, Smith BJ. Case-control analysis of ambulance, emergency room, or inpatient hospital events for epilepsy and antiepileptic drug formulation changes. Epilepsia. 2009 Mar;50(3):493-500. doi: 10.1111/j.1528-1167.2008.01703.x. Epub 2008 Jun 26. PMID 18616554
- [Background] Rascati KL, Richards KM, Johnsrud MT, Mann TA. Effects of antiepileptic drug substitutions on epileptic events requiring acute care. Pharmacotherapy. 2009 Jul;29(7):769-74. doi: 10.1592/phco.29.7.769. PMID 19558250
- [Background] Fitzgerald CL, Jacobson MP. Generic substitution of levetiracetam resulting in increased incidence of breakthrough seizures. Ann Pharmacother. 2011 May;45(5):e27. doi: 10.1345/aph.1P765. Epub 2011 Apr 26. PMID 21521860
- [Background] Bialer M, Midha KK. Generic products of antiepileptic drugs: a perspective on bioequivalence and interchangeability. Epilepsia. 2010 Jun;51(6):941-50. doi: 10.1111/j.1528-1167.2010.02573.x. Epub 2010 Apr 8. PMID 20384761
- [Background] Liow K, Barkley GL, Pollard JR, Harden CL, Bazil CW; American Academy of Neurology. Position statement on the coverage of anticonvulsant drugs for the treatment of epilepsy. Neurology. 2007 Apr 17;68(16):1249-50. doi: 10.1212/01.wnl.0000259400.30539.cc. No abstract available. PMID 17438213
- [Background] Shaw SJ, Hartman AL. The Controversy over Generic Antiepileptic Drugs. J Pediatr Pharmacol Ther. 2010 Apr;15(2):81-93. PMID 22477799
- [Background] McAuley JW, Chen AY, Elliott JO, Shneker BF. An assessment of patient and pharmacist knowledge of and attitudes toward reporting adverse drug events due to formulation switching in patients with epilepsy. Epilepsy Behav. 2009 Jan;14(1):113-7. doi: 10.1016/j.yebeh.2008.08.009. Epub 2008 Sep 26. PMID 18768168
- [Background] Ting TY, Jiang W, Lionberger R, Wong J, Jones JW, Kane MA, Krumholz A, Temple R, Polli JE. Generic lamotrigine versus brand-name Lamictal bioequivalence in patients with epilepsy: A field test of the FDA bioequivalence standard. Epilepsia. 2015 Sep;56(9):1415-24. doi: 10.1111/epi.13095. Epub 2015 Jul 23. PMID 26201987
- [Background] Stevens RE, Limsakun T, Evans G, Mason DH Jr. Controlled, multidose, pharmacokinetic evaluation of two extended-release carbamazepine formulations (Carbatrol and Tegretol-XR). J Pharm Sci. 1998 Dec;87(12):1531-4. doi: 10.1021/js980203+. PMID 10189261
- [Background] Rouits E, Burton I, Guenole E, Troenaru MM, Stockis A, Sargentini-Maier ML. Pharmacokinetics of levetiracetam XR 500mg tablets. Epilepsy Res. 2009 Apr;84(2-3):224-31. doi: 10.1016/j.eplepsyres.2009.02.001. Epub 2009 Mar 4. PMID 19264451
- [Background] Elger C, Bialer M, Falcao A, Vaz-da-Silva M, Nunes T, Almeida L, Soares-da-Silva P. Pharmacokinetics and tolerability of eslicarbazepine acetate and oxcarbazepine at steady state in healthy volunteers. Epilepsia. 2013 Aug;54(8):1453-61. doi: 10.1111/epi.12242. Epub 2013 Jun 12. PMID 23758485
- [Background] Cawello W, Bonn R. No pharmacokinetic interaction between lacosamide and valproic acid in healthy volunteers. J Clin Pharmacol. 2012 Nov;52(11):1739-48. doi: 10.1177/0091270011426875. Epub 2011 Dec 8. PMID 22162508

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1/Topiramate: Subjects received Topiramate in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Topiramate: Subjects received Topiramate in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
- Sequence 1/Lamotrigine: Subjects received Lamotrigine in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Lamotrigine: Subjects received Lamotrigine in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
- Sequence 1/Levetiracetam IR: Subjects received Levetiracetam IR in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Levetiracetam IR: Subjects received Levetiracetam IR in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
- Sequence 1/Carbamazepine ER Tablet: Subjects received Carbamazepine ER tablet in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Carbamazepine ER Tablet: Subjects received Carbamazepine ER tablet in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
- Sequence 1/Carbamazepine ER Capsule: Subjects received Carbamazepine ER capsule in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Carbamazepine ER Capsule: Subjects received Carbamazepine ER capsule in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
- Sequence 1/Zonisamide: Subjects received Zonisamide in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Zonisamide: Subjects received Zonisamide in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
- Sequence 1/Levetiracetam ER: Subjects received Levetiracetam in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Levetiracetam ER: Subjects received Levetiracetam ER in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
- Sequence 1/Valproic Acid: Subjects received Valproic acid in the sequence order 1 (TRRT).
  Test-Reference-Reference-Test
  Reference: Brand Test: Generic
- Sequence 2/Valproic Acid: Subjects received Valproic acid in the sequence order 2 (RTTR).
  Reference-Test-Test-Reference
  Reference: Brand Test: Generic
Period: Overall Study
Arm/Group | Sequence 1/Topiramate | Sequence 2/Topiramate | Sequence 1/Lamotrigine | Sequence 2/Lamotrigine | Sequence 1/Levetiracetam IR | Sequence 2/Levetiracetam IR | Sequence 1/Carbamazepine ER Tablet | Sequence 2/Carbamazepine ER Tablet | Sequence 1/Carbamazepine ER Capsule | Sequence 2/Carbamazepine ER Capsule | Sequence 1/Zonisamide | Sequence 2/Zonisamide | Sequence 1/Levetiracetam ER | Sequence 2/Levetiracetam ER | Sequence 1/Valproic Acid | Sequence 2/Valproic Acid
Started | 3 | 2 | 4 | 0 | 2 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Completed | 2 | 1 | 3 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not Completed | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PI decisions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol deviation | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received a study drug.
Groups:
- Topiramate Tablet Group: All subjects who received the Topiramate Tablet.
- Lamotrigine IR Tablet Group: All subjects who received the Lamotrigine IR Tablet.
- Lamotrigine ER Tablet Group: All subjects who received the Lamotrigine ER Tablet.
- Levetiracetam IR Tablet Group: All subjects who received the Levetiracetam IR Tablet.
- Levetiracetam ER Tablet Group: All subjects who received the Levetiracetam ER Tablet.
- Carbamazepine ER Capsule: All subjects who received the Carbamazepine ER Capsule.
- Carbamazepine ER Tablet: All subjects who received the Carbamazepine ER Tablet.
- Zonisamide Capsule Group: All subjects who received the Zonisamide Capsule.
- Valproic Acid ER Tablet Group: All subjects who received the Valproic Acid ER Tablet.
- Total: Total of all reporting groups
Arm/Group | Topiramate Tablet Group | Lamotrigine IR Tablet Group | Lamotrigine ER Tablet Group | Levetiracetam IR Tablet Group | Levetiracetam ER Tablet Group | Carbamazepine ER Capsule | Carbamazepine ER Tablet | Zonisamide Capsule Group | Valproic Acid ER Tablet Group | Total
Number analyzed (Participants) | 5 | 1 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 3 | 2 | 2 | 1 | 1 | 2 | 18
  Male | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 1 | 3 | 2 | 2 | 2 | 1 | 1 | 2 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 11
  White | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean AUC0-last_ss (Test vs. Reference)
Description: Average AUC (area under the drug plasma curve.
Time Frame: For all study drugs, time points are: predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, and 6 hr postdose. For twice-a-day regimen, additional points are:8, 10, and 12 hr postdose. For once-a-day drugs, additional times are:8, 10, 12, 16, and 24 hr postdose.
Measure: Mean (Standard Deviation); unit: micro/mL/hr
Groups:
- Topiramate Tablet: Subjects who received Topiramate for Sequence 1 and 2.
- Lamotrigine ER Tablet: Subjects who received Lamotrigine ER for Sequence 1 and 2.
- Levetiracetam IR Tablet: Subjects who received Levetiracetam IR for Sequence 1 and 2.
- Levetiracetam ER Tablet: Subjects who received Levetiracetam ER for Sequence 1 and 2.
- Carbamazepine ER Capsule: Subjects who received Carbamazepine ER Capsule for Sequence 1 and 2.
- Carbamazepine ER Tablet: Subjects who received Carbamazepine ER Tablet for Sequence 1 and 2.
- Zonisamide Capsule: Subjects who received Zonisamide for Sequence 1 and 2.
Arm/Group | Topiramate Tablet | Lamotrigine ER Tablet | Levetiracetam IR Tablet | Levetiracetam ER Tablet | Carbamazepine ER Capsule | Carbamazepine ER Tablet | Zonisamide Capsule
Number analyzed (Participants) | 5 | 3 | 3 | 2 | 1 | 1 | 1
micro/mL/hr
  Test Product | 92.884 (45.04955804) | 62.76666667 (26.51919556) | 419.97 (116.7864209) | 260.3 (169.1399421) | 114.96 (0) | 104.6 (0) | 233.16 (0)
  Reference Product | 94.456 (46.91455403) | 67.19333333 (28.83182501) | 445.2 (125.97458) | 262.305 (176.4584972) | 106.45 (0) | 115.16 (0) | 226.14 (0)

2. Primary Outcome: Mean Cmax_ss (Test vs. Reference)
Description: Average maximum drug plasma concentration;
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: microg/mL
Arm/Group | Topiramate Tablet | Lamotrigine ER Tablet | Levetiracetam IR Tablet | Levetiracetam ER Tablet | Carbamazepine ER Capsule | Carbamazepine ER Tablet | Zonisamide Capsule
Number analyzed (Participants) | 5 | 3 | 3 | 2 | 1 | 1 | 1
microg/mL
  Test Product | 9.874 (4.889389532) | 6.24 (2.327853088) | 71.02333333 (16.29206658) | 31.05 (16.64529363) | 10.95 (0) | 10.00 (0) | 12.29 (0)
  Reference Product | 9.646 (4.834328288) | 6.903333333 (2.460819647) | 69.29333333 (15.89970545) | 28.04 (17.2675476) | 9.91 (0) | 10.6 (0) | 11.68 (0)

3. Primary Outcome: Mean Cmin_ss (Test vs. Reference)
Description: Average minimum drug plasma concentration (Cmin);
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: microg/mL
Arm/Group | Topiramate Tablet | Lamotrigine ER Tablet | Levetiracetam IR Tablet | Levetiracetam ER Tablet | Carbamazepine ER Capsule | Carbamazepine ER Tablet | Zonisamide Capsule
Number analyzed (Participants) | 5 | 3 | 3 | 2 | 1 | 1 | 1
microg/mL
  Test Product | 6.326 (2.990924606) | 4.053333333 (1.569214241) | 15.45333333 (4.702981324) | 12.605 (12.21173411) | 8.56 (0) | 7.37 (0) | 8.46 (0)
  Reference Product | 6.53 (3.261203765) | 4.21 (2.343736333) | 17.45666667 (6.150612436) | 14.395 (12.40972401) | 7.66 (0) | 7.97 (0) | 8.34 (0)

4. Secondary Outcome: Number of Adverse Events
Description: summed for each anti-epileptic drug from when taking brand and generic.
Time Frame: Through the approximately 2 week period when the treatment is given.
Measure: Number; unit: events
Groups:
- Topiramate: Subjects who received Topiramate for Sequence 1 and 2.
- Lamotrigine ER: Subjects who received Lamotrigine ER for Sequence 1 and 2.
- Levetiracetam IR: Subjects who received Levetiracetam IR for Sequence 1 and 2.
- Levetiracetam ER: Subjects who received Levetiracetam ER for Sequence 1 and 2.
- Zonisamide: Subjects who received Zonisamide for Sequence 1 and 2.
- Valproic Acid: Subjects who received Valproic acid for Sequence 1 and 2.
Arm/Group | Topiramate | Lamotrigine ER | Levetiracetam IR | Levetiracetam ER | Carbamazepine ER Capsule | Zonisamide | Carbamazepine ER Tablet | Valproic Acid
Number analyzed (Participants) | 5 | 4 | 3 | 2 | 3 | 1 | 1 | 2
events | 29 | 9 | 17 | 4 | 15 | 6 | 10 | 10

5. Secondary Outcome: Number of Seizures Reported
Description: Number of seizures reported in all groups
Time Frame: Through the approximately 2 week period when the treatment is given.
Measure: Number; unit: Number of Seizures
Arm/Group | Topiramate Tablet Group | Lamotrigine IR Tablet Group | Lamotrigine ER Tablet Group | Levetiracetam IR Tablet Group | Levetiracetam ER Tablet Group | Carbamazepine ER Capsule | Carbamazepine ER Tablet | Zonisamide Capsule Group | Valproic Acid ER Tablet Group
Number analyzed (Participants) | 5 | 1 | 3 | 3 | 2 | 2 | 1 | 1 | 2
Number of Seizures
  Reference Product | 9 | 0 | 44 | 16 | 42 | 3 | 0 | 0 | 12
  Test (Generic) | 5 | 0 | 25 | 5 | 72 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 16 weeks per subject
Arm/Group | Topiramate | Lamotrigine ER | Levetiracetam IR | Levetiracetam ER | Carbamazepine ER Capsule | Zonisamide | Carbamazepine ER Tablet | Valproic Acid
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/3 | 0/2 | 0/1 | 0/1 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/3 | 0/2 | 0/1 | 0/1 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 2/3 | 2/2 | 2/3 | 1/1 | 1/1 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=5) | Lamotrigine ER (N=4) | Levetiracetam IR (N=3) | Levetiracetam ER (N=2) | Carbamazepine ER Capsule (N=3) | Zonisamide (N=1) | Carbamazepine ER Tablet (N=1) | Valproic Acid (N=2)
Worsening of aphrasia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 1 (2) | 1 (4) | 1 (1) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (3) | 1 (1) | 1 (4) | 1 (2) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (2) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swing (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Shoulder/arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The research was exploratory. The study was not a bioequivalence study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT02707965/Prot_SAP_000.pdf